CLINICAL TRIAL: NCT05669287
Title: Defining a Vascular Phenotype of Pancreatic Ductal Adenocarcinoma With CT Perfusion Using Quantitative Radiomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PERFUSION-PANC; 12034 (Other Grant/Funding Number: Dutch Cancer Society)
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-12

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: Pancreas; Pancreatic cancer; CT perfusion; Histopathology; Imaging Biomarker
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT Perfusion (Experimental): All patients will receive a baseline CT Perfusion scan. A subgroup of patients with chemotherapy treatment will receive a follow-up CT Perfusion after 3 months.
  Interventions: Diagnostic Test: CT Perfusion

INTERVENTIONS:
Diagnostic Test: CT Perfusion — CT Perfusion

SUMMARY:
With CT-perfusion(CTP) it is possible to visualize the enhancement pattern of the tumor. The perfusion CT, interleaved with a routine contrast enhanced CT (CECT) will be performed at diagnosis in all patients (goal: n=125 patients) and at the first follow-up at 3 months in patients treated with systemic therapy (goal: n=50 patients). Also, the histopathology will be collected for resected tumors to perform histopathology analysis. CTP parameters will be correlated to immunohistological findings and clinical outcome.

The main goal of the study is to create an AI-assisted method to classify patients with a vascular phenotype of pancreatic ductal adenocarcinoma (PDAC). The investigators expect that this phenotype can be used to predict overall survival and chemotherapy response.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of pancreatic cancer
* 18 years and older
* written (signed and dated) informed consent

Exclusion Criteria:

* Contra-indications to undergo CT (due to untreatable contrast allergy or renal function impairment)
* Previous treatment for pancreatic cancer
* Concomitant malignancies. Subjects with prior malignancies must be disease-free for at least 5 years
* Insufficient command of the Dutch language to be able to understand the patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Classification of vascular phenotype using CT-perfusion | Baseline
  To classify a vascular phenotype with CTP using automated perfusion analysis in patients with pancreatic ductal adenocarcinoma
Correlation of CT-perfusion features with histopathological features | Baseline, Time of Resection
  To correlate the vascular phenotype with histopathologic features (stroma and microvessel density) in patients with pancreatic ductal adenocarcinoma

SECONDARY OUTCOMES:
Association between survival and CT-perfusion features | Baseline, at 2 Years
  Automated AI analysis of survival using CT perfusion in patients with pancreatic ductal adenocarcinoma.
Prediction of chemotherapy response | Baseline, 3 Months
  Sensitivity and specificity of CT-perfusion parameters to predict chemotherapy response in patients with pancreatic ductal adenocarcinoma.
Prediction of chemotherapy response compared to RECIST | Baseline, 3 Months, 6 Months
  Sensitivity and specificity of CT-perfusion parameters to evaluate chemotherapy response in patients with pancreatic ductal adenocarcinoma, compared to RECIST 1.1 on conventional CECT.

CONTACTS AND LOCATIONS:
Overall Officials: John Hermans, MSc, MD, PhD, Principal Investigator — Radboud University Medical Center; Henkjan Huisman, MSc, PhD, Principal Investigator — Radboud University Medical Center; Lodewijk Brosens, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Hospital, Nijmegen, Gelderland, Netherlands